CLINICAL TRIAL: NCT04368260
Title: Clinical Validation of New Injection Molded Flocked Nasopharyngeal Swabs in Response to the COVID-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Amy Mathers, MD, Associate Professor, Department of Medicine, Infectious Disease, University of Virginia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSR200127
Record Dates: First submitted 2020-04-24; First posted 2020-04-29 (Actual); Results first posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: COVID19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: The primary objective of this study is to determine whether the newly designed nasopharyngeal swabs perform acceptably compared to standard swabs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Control swab (Active Comparator): FDA cleared swab
  Interventions: Device: Control swab
- Prototype swab (Experimental): Injection molded polypropylene flocked nylon NP swab
  Interventions: Device: Prototype swab

INTERVENTIONS:
Device: Control swab — FDA-cleared nasopharyngeal swab
  Arms: Control swab
Device: Prototype swab — Injection molded polypropylene flocked nylon nasopharyngeal swab
  Arms: Prototype swab

SUMMARY:
The SARS-CoV-2 pandemic has resulted in an international shortage of the nasopharyngeal (NP) swabs used to collect sample for virological testing. This shortage has become a crisis as testing capacity is growing, and threatens to become the bottleneck at University of Virginia Health System and in the Commonwealth of Virginia, as it already is in other testing centers. To resolve this crisis, a team in the Clinical Microbiology Laboratories at University of Virginia Medical Center has been working closely with biomedical engineers in the University of Virginia (UVA), School of Engineering and with high volume domestic manufacturers developing injection molded polypropylene flocked nylon NP swab.

This prototype will be tested for non-inferiority relative to existing, already validated NP swabs ("control swab") for purposes of molecular microbiology: i.e. the polymerase chain reaction (PCR) tests used for virological testing for SARS-CoV-2. Specifically, the nasopharynx of patients with Covid-19 and patients under investigation (PUI) for Covid-19, the disease caused by SARS-CoV-2, will be swabbed using a prototype swab and a control swab (the standard of care swab), and test for concordance of SARS-CoV-2. In all cases the swab will be transported in validated FDA cleared viral transport medium (VTM) as per standard operating procedure at University of Virginia Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Individuals presenting to the site for clinical care will be evaluated for clinical screening for Covid-19 testing or other respiratory infection testing.
* Individuals felt identified clinically as needing Covid-19 testing may be approached for study participation.
* Individuals already under clinical care that have tested positive for Covid-19 will be approached for study participation.
* Volunteer health care workers who have approached the Principal Investigator

Exclusion Criteria:

* Known thrombocytopenia of <50,000 platelets/μl (risk of mild bleeding).
* Individuals presenting with an anatomically altered nasal cavity.
* Pregnant (self-reported)
* No other patients will be specifically excluded.

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Mathers, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) that underlie results in a publication will be shared.
Time Frame: Starting 6 months after publication
Access Criteria: Requests to made to Principal Investigator

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: 40 subjects with either presumed positive COVID-19 status or presumed negative COVID-19 status were included in this study. Control and prototype nasopharyngeal swabs were collected from each subject.
Period: Overall Study
Arm/Group | All Study Participants
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 40
Presumed COVID-19 Status [Count of Participants; unit: Participants]
  Presumed COVID-19 Positive | 20
  Presumed COVID-19 Negative | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects for Which the Prototype Swab and the Control Swab Provide the Same COVID-19 PCR Result
Description: Both the prototype and control nasopharyngeal swabs will be utilized in each subject. The rate of agreement between the swabs will be determined by the number of subjects for which both swabs provide the same COVID-19 PCR result.
Time Frame: at time of enrollment
Measure: Number; unit: participants
Arm/Group | Control Swab | Prototype Swab
Number analyzed (Participants) | 40 | 40
participants
  Positive Sample | 18 | 17
  Negative Sample | 22 | 23

ADVERSE EVENTS:
Time Frame: 1 Day
Arm/Group | Control Swab | Prototype Swab
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/60/NCT04368260/Prot_SAP_000.pdf